CLINICAL TRIAL: NCT05590286
Title: A RCT of the Efficacy of Vonoprazan 20mg QD Combined With Amoxicillin 750mg QID in the Treatment of Helicobacter Pylori Infection
Brief Title: A RCT of the Efficacy of Vonoprazan 20mg QD in the Treatment of Helicobacter Pylori Infection
Acronym: VATH-1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, ZhangXiaofeng, chief physician, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-183
Record Dates: First submitted 2022-10-19; First posted 2022-10-21 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Vonoprazan; Helicobacter Pylori Infection; Proton Pump Inhibitor
Keywords: vonoprazan; Helicobacter Pylori; Proton pump inhibitor
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vonoprazan 20mg QD (Experimental): Vonoprazan 20 mg, tablets, orally, qd given in combination with amoxicillin 750mg capsules, orally, qid for up to 2 weeks.
  Interventions: Drug: Vonoprazan Tablets; Drug: Amoxicillin Capsules
- esomeprazole 20 mg BID (Active Comparator): esomeprazole 20 mg, tablets, orally, bid given in combination with amoxicillin 1000mg，clarithromycin 500mg bid，colloidal bismuth pectin 200mg bid for up to 2 weeks.
  OR esomeprazole 20 mg, tablets, orally, bis in die given in combination with amoxicillin 750mg capsules, orally, quarter die for up to 2 weeks.
  Interventions: Drug: Amoxicillin Capsules; Drug: Esomeprazole

INTERVENTIONS:
Drug: Vonoprazan Tablets — Vonoprazan 20 mg, tablets, orally，QD
  Arms: vonoprazan 20mg QD
Drug: Amoxicillin Capsules — Amoxicillin 750mg, Capsules ,orally，QID
Drug: Esomeprazole — Esomeprazole 20mg, Capsules ,orally，BID
  Arms: esomeprazole 20 mg BID

SUMMARY:
The treatment of helicobacter pylori is very important. The routine treatment is quadruple therapy. In recent years, double therapy has appeared and the curative effect is fair. However, antacid generally uses proton pump inhibitor. The proton pump inhibitor needs double dose to achieve good antacid curative effect. The effect of vonoprazan used for inhibiting gastric acid is better than proton pump inhibitor. At present, many studies use vonoprazan instead of common proton pump inhibitor, but almost all use double dose of vonoprazan. In the previous study, we found that the effect of double dose of proton pump inhibitor can be achieved with 20mg QD of vonoprazan. Therefore, in this study, 20mg QD of vonoprazan was used to replace the double dose of proton pump inhibitor to observe the antibacterial effect of vonoprazan on Helicobacter pylori.

DETAILED DESCRIPTION:
The treatment of helicobacter pylori is very important. The routine treatment is quadruple therapy. In recent years, double therapy has appeared and the curative effect is fair. However, antacid generally uses proton pump inhibitor. The proton pump inhibitor needs double dose to achieve good antacid curative effect. The effect of vonoprazan used for inhibiting gastric acid is better than proton pump inhibitor. At present, many studies use vonoprazan instead of common proton pump inhibitor, but almost all use double dose of vonoprazan. In the previous study, we found that the effect of double dose of proton pump inhibitor can be achieved with 20mg QD of vonoprazan. Therefore, in this study, 20mg QD of vonoprazan was used to replace the double dose of proton pump inhibitor to observe the antibacterial effect of vonoprazan on Helicobacter pylori.

ELIGIBILITY:
Patients aged ≥18 years with Hp-positive first sterilization were included in this study. Before treatment, the existence of Helicobacter pylori can be confirmed by one or more of the following methods: rapid urease test, Hp culture, 13C urea breath test, 14C urea breath test and stool Hp antigen test.

The main exclusion criteria include acute upper gastrointestinal bleeding, active gastric or duodenal ulcer, acute gastric or duodenal mucosal lesions, previous eradication treatment of Helicobacter pylori, penicillin/furazolidone allergy, surgery that may affect gastric acid secretion (upper gastrointestinal resection or vagotomy), Zollinger-Ellison syndrome or other hypergastric acid secretion diseases, severe neurological, cardiovascular, pulmonary, liver, renal, metabolic, gastrointestinal, urological, etc. Any fertile woman must use proper contraception. All subjects provided written informed consent before participating in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Helicobacter Pylori Positive (HP+) Participants With Successful HP Eradication at Week 4 Post-Treatment | Week 4 post-treatment
  HP infection status will be determined by ^13C Urea Breath Test (^13C-UBT). The urea breath test is used to detect infection with HP, a bacteria associated with stomach ulcers, by testing individual breath samples in a central laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou first people's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No